CLINICAL TRIAL: NCT00597675
Title: Oral Immunotherapy for Peanut Allergy (2nd Generation PMIT Collaboration With Arkansas Children's)
Brief Title: Oral Immunotherapy for Peanut Allergy (PMIT)
Acronym: PMIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00000163
Record Dates: First submitted 2008-01-04; First posted 2008-01-18 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2017-03

CONDITIONS: Food Hypersensitivity
Keywords: Peanut allergy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Oat flour ingested daily as a placebo
  Interventions: Biological: Placebo
- Peanut OIT (Active Comparator): Peanut flour ingested daily as oral mucosal immunotherapy
  Interventions: Biological: Peanut OIT

INTERVENTIONS:
Biological: Peanut OIT — Defatted peanut flour ingested daily as oral mucosal immunotherapy
  Arms: Peanut OIT
Biological: Placebo — Oat flour matched by weight and consistency that is ingested daily as a placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if mucosal peanut immunotherapy will make subjects who have peanut allergy less allergic and induce changes in their immune system.

DETAILED DESCRIPTION:
Peanut allergy is known to cause severe anaphylactic reactions. Compared with other food allergies it tends to be more persistent and also its prevalence seems to be rising. Currently there is no proven treatment other than strict avoidance. We are attempting to decrease the risk of anaphylaxis on accidental ingestion by desensitizing subjects to peanut using peanut oral mucosal immunotherapy (OIT). We are also studying the effect of peanut OIT on the peanut specific immune response to determine if tolerance to peanut protein will develop. Children ages 1 to 18 with peanut allergy will be randomized to peanut OIT or placebo. Subjects will undergo a modified rush immunotherapy on the first day and then increase the doses at least every two weeks up to a maintenance dose of 4 grams (equivalent to about 13 peanuts). Doses will be taken daily at home except for dose increases which will be done on the research unit. Subjects will undergo a double-blind, placebo-controlled food challenge (DBPCFC) after 12 months and then be unblinded. Placebo subjects will cross over to open-label peanut OIT and undergo an identical buildup schedule up to 12 months. All subjects will then complete at least 36 months of peanut OIT therapy after which once skin prick (<5 mm) and IgE (<15 kU/L) criteria are met, they will then complete the end of study DBPCFC. Dosing will continue up to a maximum of 60 months after which even if criteria are not met, the subject will undergo the end of study DBPCFC. Outcome variables of interest include response to DBPCFC, skin prick testing, peanut specific IgE, and adverse events. These results will be compared between the start and end of peanut OIT using appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject between 1 and 18 years of age
* EITHER history of significant clinical symptoms occurring within 60 minutes after ingesting peanuts greater than 6 months ago AND peanut specific IgE >15 kU/L
* OR history of significant clinical symptoms occurring within 60 minutes after ingesting peanuts within the past 6 months AND peanut specific IgE > 7 kU/L
* A family that will be able to be compliant with all study visits
* All females of child bearing age must be using appropriate birth control

Exclusion Criteria:

* Subjects with a history of severe, anaphylaxis to peanut
* Medical history that would prevent a double blind placebo controlled oral food challenge (DBPCFC/OFC) to peanut
* Unable to cooperate with challenge procedures or unable to be reached by telephone for follow-up
* Diagnosed oat allergy
* Pregnancy or lactation

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arvil W Burks, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oat flour taken daily as a placebo
- Peanut OIT: Peanut flour ingested daily as active OIT treatment
Period: Blinded Phase
Arm/Group | Placebo | Peanut OIT
Started | 4 | 6
Completed | 2 | 5
Not Completed | 2 | 1
Period: Open Label Phase
Arm/Group | Placebo | Peanut OIT
Started | 2 (Patients previously on placebo were crossed over onto open label peanut OIT) | 5
Completed | 2 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Peanut OIT | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Full Range); unit: years] | 5.8 [4.8 to 6.9] | 5.2 [3.6 to 7.0] | 5.4 [3.6 to 7.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Amount of Peanut Protein Ingested Before An Allergic Reaction is Observed During the Double-blind, Placebo Controlled Food Challenge (DBPCFC) After Completing Treatment With Peanut OIT.
Description: After completing the peanut OIT protocol (defined as treatment with peanut OIT for at least 36-months AND a peanut-specific IgE >2 and <15 AND skin prick test is <5 mm OR a maximum of 60 months of treatment), the reaction threshold for subjects is assessed by a DBPCFC. This involves eating small increasing doses of peanut protein in a blinded fashion up to a cumulative total of 5000 mg. An identical food challenge is also performed with oat flour as a placebo. The cumulative amount of peanut protein ingested prior to the dose that causes a reaction requiring treatment is reported as the reaction threshold.
Time Frame: 36-60 months
Measure: Median (Full Range); unit: mg of peanut protein
Groups:
- Open Label Peanut OIT: All subjects on active treatment after placebo subjects have been crossed over to open label treatment
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 7
mg of peanut protein | 5000 [3750 to 5000]

2. Secondary Outcome: The Amount of Peanut Protein Ingested Before An Allergic Reaction is Observed During the Double-blind, Placebo Controlled Food Challenge (DBPCFC) After Completing 12 Months of Blinded Peanut OIT or Placebo Treatment.
Description: After 12 months of blinded Peanut OIT treatment, the reaction threshold for subjects is assessed by a DBPCFC. This involves eating small increasing doses of peanut protein in a blinded fashion up to a cumulative total of 4710 mg. An identical food challenge is also performed with oat flour as a placebo. The cumulative amount of peanut protein ingested prior to the dose that causes a reaction requiring treatment is reported as the reaction threshold.
Time Frame: 12 months
Measure: Median (Full Range); unit: mg of peanut protein
Arm/Group | Placebo | Peanut OIT
Number analyzed (Participants) | 4 | 5
mg of peanut protein | 123 [35 to 210] | 4710 [4710 to 4710]

3. Secondary Outcome: The Change From Baseline Through the End of Peanut OIT Treatment in Wheal Size Diameter Following Peanut Skin Prick Testing
Description: Skin prick testing is performed by scratching the skin with a small amount of peanut and observing for redness and a raised bump called a wheal. The diameter of the wheal is measured with a ruler in mm and recorded as a measure of peanut-specific IgE and mast cell reactivity in an allergic subject. A decrease in wheal size after treatment would represent suppression of the allergic response.
Time Frame: Baseline to end of open label phase treatment (36-60 months)
Measure: Median (Full Range); unit: mm
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 7
mm | -4.5 [-21 to 3.3]

4. Secondary Outcome: The Change From Baseline Through the End of Peanut OIT Treatment in Peanut-specific IgE in the Blood
Description: Peanut specific IgE on the surface of mast cells and basophils releases histamine when exposed to peanut causing symptoms of allergy. Free-floating peanut-specific IgE is measured from serum in the blood by an immunoCAP machine and reported in kU/L. A lower level of peanut-specific IgE could suggest a decrease in the probability of reaction for a subject who is exposed to peanut.
Time Frame: Baseline to end of open label phase treatment (36-60 months)
Measure: Median (Full Range); unit: kU/L
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 7
kU/L | -187 [-658.5 to -19.4]

5. Secondary Outcome: The Change From Baseline Through the End of Peanut OIT Treatment in Peanut-specific IgG4 in the Blood.
Description: Peanut specific IgG4 is thought to have a protective effect for a subject when exposed to peanut possibly by interfering with IgE. Peanut-specific IgG4 is measured from serum in the blood by an immunoCAP machine and reported in mg/dL. A higher level of peanut-specific IgG4 could suggest a decrease in the probability of reaction for a subject who is exposed to peanut.
Time Frame: Baseline to end of open label phase treatment (36-60 months)
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 7
mg/dL | 6.6 [0.7 to 95.5]

ADVERSE EVENTS:
Time Frame: During the initial 12 months of the study, subjects were blinded and adverse events were reported separately for treatment and placebo groups. During the open label phase of treatment, adverse events were reported for the entire cohort. For subjects on active therapy, open-label was from after unblinding at 12 months through 36-60 months. For subjects on placebo, open-label was from crossing over to peanut OIT at time 0 through 36-60 months of active treatment.
Groups:
- Open Label Phase-Peanut OIT: All subjects receiving open-label peanut OIT from the point of unblinding through the end of the treatment phase.
- Blinded Phase-Placebo: Patients receiving oat flour as a placebo during the initial 12 months of therapy.
- Blinded Phase-Peanut OIT: Patients receiving peanut flour as active OIT during the initial 12 months of therapy.
Arm/Group | Open Label Phase-Peanut OIT | Blinded Phase-Placebo | Blinded Phase-Peanut OIT
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 6/9 | 4/4 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Phase-Peanut OIT (N=9) | Blinded Phase-Placebo (N=4) | Blinded Phase-Peanut OIT (N=6)
Vomiting (Gastrointestinal disorders) | 2 | 1 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Erythematous rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Oropharyngeal itching (Gastrointestinal disorders) | 2 | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Itchy nose (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin itch (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Lip or eye swelling (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Eye itch (Eye disorders) | 2 | 1 | 1
Eye tearing (Eye disorders) | 0 | 1 | 0
Hives (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No